CLINICAL TRIAL: NCT02083172
Title: Evaluating Agreement Between USCOM and 2D-echocardiographic Hemodynamic Measurements in Pediatric Patients
Brief Title: Comparing USCOM and Echocardiographic Hemodynamic Measurements in Children (CUE Study)
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Karen Choong, Associate professor, Departments of Pediatrics and Critical Care, McMaster University
Other Study IDs: 13-658
Record Dates: First submitted 2013-11-25; First posted 2014-03-11 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2015-11

CONDITIONS: Hemodynamically Stable; Critical Illness
Keywords: USCOM (UltraSound Cardiac Output Monitor); 2D echocardiography; agreement; pediatrics
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Hemodynamically stable patients: Hemodynamically stable patients will be defined as patients with normal hemodynamic profile as evidenced by normal age-determined vital signs and normal perfusion.
  Interventions: Device: Ultrasound Cardiac Output Monitor and 2 D-Echo
- Hemodynamically unstable patients: Hemodynamically unstable patients will be defined as patients who are admitted to the Pediatric Critical Care Unit (PCCU), in whom there is a clinical diagnosis of shock as evidenced by signs and symptoms of hypoperfusion, requiring fluid resuscitation and/or inotropic support.
  Interventions: Device: Ultrasound Cardiac Output Monitor and 2 D-Echo
- Mechanically ventilated patients: Patients requiring mechanical ventilation
  Interventions: Device: Ultrasound Cardiac Output Monitor and 2 D-Echo

INTERVENTIONS:
Device: Ultrasound Cardiac Output Monitor and 2 D-Echo — Hemodynamic measurements obtained by 2D-Echo and USCOM will be compared.
  Other Names: USCOM

SUMMARY:
The primary objective of this study is to evaluate the agreement between hemodynamic measurements obtained using the Ultrasound Cardiac Output Monitor (USCOM®; USCOM Ltd., Sydney, Australia), and reference standards as determined by 2 Dimensional echocardiography (2D-echo) measurements in a group of hemodynamically stable and unstable pediatric patients.

DETAILED DESCRIPTION:
2D-echo is the standard-of-care tool for non-invasive hemodynamic assessments in children. The use of 2D-echo requires highly trained personnel, and assessments may take anywhere between 30-45 minutes. The feasibility of real time hemodynamic assessments is therefore limited with 2D-echo. USCOM has been introduced as a non-invasive bedside hemodynamic monitoring tool that utilizes continuous-wave Doppler ultrasound. As USCOM is easily portable, and measurements take only several minutes and can be conducted by trained physicians or nurses, it has become an attractive method of real time hemodynamic monitoring of unstable patients. While USCOM validation studies have been conducted in adult, neonatal and pediatric populations, the following concerns have been raised: a) Pediatric data on the agreement between USCOM and other standard methods of CO measurement (i.e. 2D-echo, pulmonary artery catheterization) are conflicting with some studies reporting acceptable agreement, while others report poor agreement ; b) USCOM validation and agreement studies were previously conducted in primarily hemodynamically stable populations. Its performance in hemodynamically unstable and mechanically ventilated patients has not been studied to date in the pediatric population.USCOM is currently being promoted as a real-time tool for assessing hemodynamic status, and directing the care of unstable children without adequate evidence. Therefore, this study is essential to inform the validity of USCOM and whether it can or should be used when 2D-echo for real time hemodynamic monitoring in children is not feasible or available.

ELIGIBILITY:
Inclusion Criteria:

* Age under 18 years
* Patient fulfills clinical criteria for either study cohort
* Most Responsible Physician has ordered an ECHO study on the patient
* Written informed consent by parents/legal guardian/substitute decision maker, and assent where appropriate
* Patients with normal cardiac structure, no pre-existing primary cardiovascular disease or hemodynamically insignificant shunt lesions (i.e. hemodynamically insignificant Atrial Septal Defect/Patent Foramen Oval and Ventricular Septal Defect

Exclusion Criteria:

* Age ≥ 18 years
* Premature infants (born <37 weeks gestation) admitted to the Neonatal Intensive Care Unit
* Known co-existing primary cardiac anomalies (i.e. aortic or pulmonary valve stenosis or regurgitation, Aortic Valve regurgitation, shunt lesions save for those mentioned above, and pericardial effusion)
* Prior enrollment in study

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1. The hemodynamically stable group: will be screened from pediatric in-patients on McMaster Children's Hospital general pediatric wards and those scheduled for elective 2D-echo through cardiology and sedation clinic.
  2. The hemodynamically unstable patients and 3. those requiring mechanical ventilation will be screened from McMaster Children's Hospital Pediatric Critical Care Unit.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Agreement in hemodynamic measurements obtained by USCOM and 2D-Echo respectively, in hemodynamically stable children | Within 30 minutes of first measurement method
  Hemodynamic measurements are include cardiac output (CO), Stroke Volume (SV),Aortic cross sectional area (Ao CSA), Preload (SVV%) Inferior Vena cava Collapsibility index (IVC), Inotropy (SMI) and (EF)

SECONDARY OUTCOMES:
Agreement in hemodynamic measurements obtained by USCOM and 2D-Echo, in hemodynamically unstable children, and children receiving positive pressure ventilation respectively | Within 30 minutes of first measurement method
  Hemodynamic measurements are include Cardiac Output (CO), Stroke Volume(SV), Preload (SVV%) and IVC collapsibility Index, Inotropy

CONTACTS AND LOCATIONS:
Overall Officials: Karen Choong, MD,BCh,MSc, Study Chair — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Background] Odetola FO, Gebremariam A, Freed GL. Patient and hospital correlates of clinical outcomes and resource utilization in severe pediatric sepsis. Pediatrics. 2007 Mar;119(3):487-94. doi: 10.1542/peds.2006-2353. PMID 17332201
- [Background] Parrillo JE, Parker MM, Natanson C, Suffredini AF, Danner RL, Cunnion RE, Ognibene FP. Septic shock in humans. Advances in the understanding of pathogenesis, cardiovascular dysfunction, and therapy. Ann Intern Med. 1990 Aug 1;113(3):227-42. doi: 10.7326/0003-4819-113-3-227. PMID 2197912
- [Background] Zanotti-Cavazzoni SL, Hollenberg SM. Cardiac dysfunction in severe sepsis and septic shock. Curr Opin Crit Care. 2009 Oct;15(5):392-7. doi: 10.1097/MCC.0b013e3283307a4e. PMID 19633546
- [Background] Kumar A, Haery C, Parrillo JE. Myocardial dysfunction in septic shock. Crit Care Clin. 2000 Apr;16(2):251-87. doi: 10.1016/s0749-0704(05)70110-x. PMID 10768082
- [Background] Brierley J, Carcillo JA, Choong K, Cornell T, Decaen A, Deymann A, Doctor A, Davis A, Duff J, Dugas MA, Duncan A, Evans B, Feldman J, Felmet K, Fisher G, Frankel L, Jeffries H, Greenwald B, Gutierrez J, Hall M, Han YY, Hanson J, Hazelzet J, Hernan L, Kiff J, Kissoon N, Kon A, Irazuzta J, Lin J, Lorts A, Mariscalco M, Mehta R, Nadel S, Nguyen T, Nicholson C, Peters M, Okhuysen-Cawley R, Poulton T, Relves M, Rodriguez A, Rozenfeld R, Schnitzler E, Shanley T, Kache S, Skippen P, Torres A, von Dessauer B, Weingarten J, Yeh T, Zaritsky A, Stojadinovic B, Zimmerman J, Zuckerberg A. Clinical practice parameters for hemodynamic support of pediatric and neonatal septic shock: 2007 update from the American College of Critical Care Medicine. Crit Care Med. 2009 Feb;37(2):666-88. doi: 10.1097/CCM.0b013e31819323c6. PMID 19325359
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Kern JW, Shoemaker WC. Meta-analysis of hemodynamic optimization in high-risk patients. Crit Care Med. 2002 Aug;30(8):1686-92. doi: 10.1097/00003246-200208000-00002. PMID 12163777
- [Background] Lapostolle F, Petrovic T, Catineau J, Lenoir G, Adnet F. Training emergency physicians to perform out-of-hospital ultrasonography. Am J Emerg Med. 2005 Jul;23(4):572. doi: 10.1016/j.ajem.2005.01.008. No abstract available. PMID 16032640
- [Background] Stewart GM, Nguyen HB, Kim TY, Jauregui J, Hayes SR, Corbett S. Inter-rater reliability for noninvasive measurement of cardiac function in children. Pediatr Emerg Care. 2008 Jul;24(7):433-7. doi: 10.1097/PEC.0b013e31817de143. PMID 18580818
- [Background] Meyer S, Todd D, Shadboldt B. Assessment of portable continuous wave Doppler ultrasound (ultrasonic cardiac output monitor) for cardiac output measurements in neonates. J Paediatr Child Health. 2009 Jul-Aug;45(7-8):464-8. doi: 10.1111/j.1440-1754.2009.01535.x. PMID 19712182
- [Background] Critchley LA, Peng ZY, Fok BS, Lee A, Phillips RA. Testing the reliability of a new ultrasonic cardiac output monitor, the USCOM, by using aortic flowprobes in anesthetized dogs. Anesth Analg. 2005 Mar;100(3):748-753. doi: 10.1213/01.ANE.0000144774.42408.05. PMID 15728064
- [Background] Su BC, Yu HP, Yang MW, Lin CC, Kao MC, Chang CH, Lee WC. Reliability of a new ultrasonic cardiac output monitor in recipients of living donor liver transplantation. Liver Transpl. 2008 Jul;14(7):1029-37. doi: 10.1002/lt.21461. PMID 18581505
- [Background] He SR, Zhang C, Liu YM, Sun YX, Zhuang J, Chen JM, Madigan VM, Smith BE, Sun X. Accuracy of the ultrasonic cardiac output monitor in healthy term neonates during postnatal circulatory adaptation. Chin Med J (Engl). 2011 Aug;124(15):2284-9. PMID 21933558
- [Background] Brierley J, Peters MJ. Distinct hemodynamic patterns of septic shock at presentation to pediatric intensive care. Pediatrics. 2008 Oct;122(4):752-9. doi: 10.1542/peds.2007-1979. PMID 18829798
- [Background] van Lelyveld-Haas LE, van Zanten AR, Borm GF, Tjan DH. Clinical validation of the non-invasive cardiac output monitor USCOM-1A in critically ill patients. Eur J Anaesthesiol. 2008 Nov;25(11):917-24. doi: 10.1017/S0265021508004882. Epub 2008 Jul 24. PMID 18652712
- [Background] Tan HL, Pinder M, Parsons R, Roberts B, van Heerden PV. Clinical evaluation of USCOM ultrasonic cardiac output monitor in cardiac surgical patients in intensive care unit. Br J Anaesth. 2005 Mar;94(3):287-91. doi: 10.1093/bja/aei054. Epub 2005 Jan 14. PMID 15653709
- [Background] Chand R, Mehta Y, Trehan N. Cardiac output estimation with a new Doppler device after off-pump coronary artery bypass surgery. J Cardiothorac Vasc Anesth. 2006 Jun;20(3):315-9. doi: 10.1053/j.jvca.2005.05.024. Epub 2006 Jan 18. PMID 16750729
- [Background] Deep A, Goonasekera CD, Wang Y, Brierley J. Evolution of haemodynamics and outcome of fluid-refractory septic shock in children. Intensive Care Med. 2013 Sep;39(9):1602-9. doi: 10.1007/s00134-013-3003-z. Epub 2013 Jun 28. PMID 23812341
- [Background] Dellinger RP, Levy MM, Carlet JM, Bion J, Parker MM, Jaeschke R, Reinhart K, Angus DC, Brun-Buisson C, Beale R, Calandra T, Dhainaut JF, Gerlach H, Harvey M, Marini JJ, Marshall J, Ranieri M, Ramsay G, Sevransky J, Thompson BT, Townsend S, Vender JS, Zimmerman JL, Vincent JL. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock: 2008. Intensive Care Med. 2008 Jan;34(1):17-60. doi: 10.1007/s00134-007-0934-2. Epub 2007 Dec 4. PMID 18058085
- [Background] Zheng ML, Sun X, Zhong J, He SR, Pan W, Pang CC, Sun YX, Liu YM. [Clinical study of neonatal cardiac output measurement methods]. Zhonghua Er Ke Za Zhi. 2013 Jan;51(1):58-63. Chinese. PMID 23527933
- [Background] Wongsirimetheekul T, Khositseth A, Lerbunrian R. (2013). Noninvasive cardiac output assessment in critically ill pediatric patients [poster]. Am J Respir Crit Care Med 187: A3686.
- [Background] Lichtenthal PR, Sloniger JA, Copeland JG. (2007) USCOM non-invasive Doppler cardiac output: Are measurements accurate in infants and children? Anesthesiology 107: A1528.
- [Background] Eguchi JH,Mathur M,Larsen R,et al.Ultrasound cardiac output monitor measurement in pediatric cardiac transplant patients.J Heart Lung Transplant,2007,26 (2):S136.
- [Background] Lichtenthal PR, Phillips RA, Sloniger JA, et al. (2006) USCOM non-invasive Doppler: Are cardiac output measurements accurate in both infants and adults? Anesthesiology 105: A466
- [Background] Phillips RA, Paradisis M, Evans NJ, et al. (2006) Validation of USCOM CO measurements in preterm neonates by comparison with echocardiography. Crit Care Med 10(S1): 144-343
- [Background] Patel N, Dodsworth M, Mills JF. Cardiac output measurement in newborn infants using the ultrasonic cardiac output monitor: an assessment of agreement with conventional echocardiography, repeatability and new user experience. Arch Dis Child Fetal Neonatal Ed. 2011 May;96(3):F206-11. doi: 10.1136/adc.2009.170704. Epub 2010 Jul 6. PMID 20605971
- [Background] Nguyen HB, Banta DP, Stewart G, Kim T, Bansal R, Anholm J, Wittlake WA, Corbett SW. Cardiac index measurements by transcutaneous Doppler ultrasound and transthoracic echocardiography in adult and pediatric emergency patients. J Clin Monit Comput. 2010 Jun;24(3):237-47. doi: 10.1007/s10877-010-9240-6. Epub 2010 Jun 20. PMID 20563629
- [Background] Knirsch W, Kretschmar O, Tomaske M, Stutz K, Nagdyman N, Balmer C, Schmitz A, Bettex D, Berger F, Bauersfeld U, Weiss M. Cardiac output measurement in children: comparison of the Ultrasound Cardiac Output Monitor with thermodilution cardiac output measurement. Intensive Care Med. 2008 Jun;34(6):1060-4. doi: 10.1007/s00134-008-1030-y. Epub 2008 Feb 23. PMID 18297271
- [Background] Jain S, Allins A, Salim A, Vafa A, Wilson MT, Margulies DR. Noninvasive Doppler ultrasonography for assessing cardiac function: can it replace the Swan-Ganz catheter? Am J Surg. 2008 Dec;196(6):961-7; discussion 967-8. doi: 10.1016/j.amjsurg.2008.07.039. PMID 19095116
- [Background] Lang RM, Bierig M, Devereux RB, Flachskampf FA, Foster E, Pellikka PA, Picard MH, Roman MJ, Seward J, Shanewise JS, Solomon SD, Spencer KT, Sutton MS, Stewart WJ; Chamber Quantification Writing Group; American Society of Echocardiography's Guidelines and Standards Committee; European Association of Echocardiography. Recommendations for chamber quantification: a report from the American Society of Echocardiography's Guidelines and Standards Committee and the Chamber Quantification Writing Group, developed in conjunction with the European Association of Echocardiography, a branch of the European Society of Cardiology. J Am Soc Echocardiogr. 2005 Dec;18(12):1440-63. doi: 10.1016/j.echo.2005.10.005. No abstract available. PMID 16376782
- [Background] Krause I, Birk E, Davidovits M, Cleper R, Blieden L, Pinhas L, Gamzo Z, Eisenstein B. Inferior vena cava diameter: a useful method for estimation of fluid status in children on haemodialysis. Nephrol Dial Transplant. 2001 Jun;16(6):1203-6. doi: 10.1093/ndt/16.6.1203. PMID 11390721
- [Background] Kosiak W, Swieton D, Piskunowicz M. Sonographic inferior vena cava/aorta diameter index, a new approach to the body fluid status assessment in children and young adults in emergency ultrasound--preliminary study. Am J Emerg Med. 2008 Mar;26(3):320-5. doi: 10.1016/j.ajem.2007.07.012. PMID 18358944
- [Background] Chen L, Kim Y, Santucci KA. Use of ultrasound measurement of the inferior vena cava diameter as an objective tool in the assessment of children with clinical dehydration. Acad Emerg Med. 2007 Oct;14(10):841-5. doi: 10.1197/j.aem.2007.06.040. PMID 17898246
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Meyer S, Todd D, Wright I, Gortner L, Reynolds G. Review article: Non-invasive assessment of cardiac output with portable continuous-wave Doppler ultrasound. Emerg Med Australas. 2008 Jun;20(3):201-8. doi: 10.1111/j.1742-6723.2008.01078.x. Epub 2008 Apr 9. PMID 18400002
- [Background] Levy JA, Noble VE. Bedside ultrasound in pediatric emergency medicine. Pediatrics. 2008 May;121(5):e1404-12. doi: 10.1542/peds.2007-1816. PMID 18450883
- [Background] Barnett SB, Ter Haar GR, Ziskin MC, Rott HD, Duck FA, Maeda K. International recommendations and guidelines for the safe use of diagnostic ultrasound in medicine. Ultrasound Med Biol. 2000 Mar;26(3):355-66. doi: 10.1016/s0301-5629(00)00204-0. PMID 10773365
- [Background] Hershkovitz R, Sheiner E, Mazor M. Ultrasound in obstetrics: a review of safety. Eur J Obstet Gynecol Reprod Biol. 2002 Feb 10;101(1):15-8. doi: 10.1016/s0301-2115(01)00469-9. PMID 11803093
- [Background] Schratz LM, Meyer RA, Schwartz DC. Serial intracoronary ultrasound in children: feasibility, reproducibility, limitations, and safety. J Am Soc Echocardiogr. 2002 Aug;15(8):782-90. doi: 10.1067/mje.2002.119911. PMID 12174347
- [Background] Mosteller RD. Simplified calculation of body-surface area. N Engl J Med. 1987 Oct 22;317(17):1098. doi: 10.1056/NEJM198710223171717. No abstract available. PMID 3657876